CLINICAL TRIAL: NCT07320183
Title: Effect of a Dietary Supplement Containing EGCG, Folic Acid, Vitamin B12 and Hyaluronic Acid in Supporting Male Genital Balance in Subjects Exposed to HPV Risk
Acronym: PERVI-M
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Lo.Li.Pharma s.r.l (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 8299
Record Dates: First submitted 2025-12-22; First posted 2026-01-06 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: HPV - Anogenital Human Papilloma Virus Infection; Infertilities
Keywords: HPV- infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients taking Pervistop (Experimental): 24 couples in which both partners will receive a supplement containing EGCG (200 mg), vitamin B12 (1 mg), hyaluronic acid (50 mg), and folic acid (400 μg), one tablet daily orally for 6 month
  Interventions: Dietary Supplement: pervistop
- Patients no taking Pervistop (No Intervention): 24 couples with no supplementation.

INTERVENTIONS:
Dietary Supplement: pervistop — combination of EGCG, vitamin B12, hyaluronic acid, and folic acid
  Arms: Patients taking Pervistop

SUMMARY:
Pilot interventional study aimed at evaluating the effect of a dietary supplement containing EGCG, vitamin B12, hyaluronic acid, and folic acid on the maintenance of physiological balance of the genital mucosa and natural defenses of the male genital tract, as well as on the maintenance of HPV-DNA test negativity, in subjects undergoing natural procreation pathways. The study will also assess the potential support of sperm parameters, reproductive well-being of the couple, and the reduction of risk factors associated with HPV transmission to the female partner. A total of 34 HPV-positive couples attending the Istituto Scientifico Internazionale "Paolo VI" of the Policlinico A. Gemelli will be enrolled and randomized into two groups: 17 couples in the intervention group, in which the male partner will receive the supplement (EGCG 200 mg, vitamin B12 1 mg, hyaluronic acid 50 mg, folic acid 400 μg, one tablet daily for 6 months), and 17 couples in the control group with no supplementation.

DETAILED DESCRIPTION:
This pilot, randomized interventional study aims to assess the effect of a dietary supplement containing epigallocatechin gallate (EGCG), vitamin B12, hyaluronic acid, and folic acid on the maintenance of physiological balance and natural defenses of the male genital tract in men with HPV infection attending natural procreation centers. The study also seeks to evaluate whether supplementation may support sperm quality, improve reproductive well-being of participating couples, and reduce risk factors associated with HPV transmission to the female partner.

A total of 48 couples (96 participants) will be enrolled at the Istituto Scientifico Internazionale "Paolo VI" of the Policlinico A. Gemelli. Eligible couples, characterized by an HPV-positive male partner and an HPV-negative female partner, will be randomized into two groups: a supplement group, in which both partners will receive oral supplementation with EGCG (200 mg), vitamin B12 (1 mg), hyaluronic acid (50 mg), and folic acid (400 μg) once daily for 6 months, and a control group receiving no supplementation. Randomization will be performed using a computer-generated list.

The primary endpoint is the proportion of male participants achieving a negative HPV DNA test at the end of the 6-month intervention period. Secondary endpoints include changes in sperm quality parameters assessed by semen analysis according to WHO 2021 guidelines, measures of reproductive outcomes such as fertility potential and achievement of pregnancy, and maintenance of genital mucosal health, including absence of infections or recurrences and reduced risk of HPV transmission. HPV genotyping will be assessed by PCR on urethral swab samples. The overall study duration is expected to be 18 months following ethics committee approval.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Couple seeking pregnancy
* Male partner aged 25-65 years
* HPV DNA test indicating active HPV infection in the male partner
* HPV DNA test indicating negativity for HPV infection in the female partner

Exclusion Criteria:

* Concomitant diseases causing immunosuppression
* Treatment with immunomodulatory therapies
* Use of EGCG or other green tea extracts

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 96 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Negative HPV-DNA test | 6 months
  Proportion of participants with a negative HPV DNA test at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Domenico Milardi, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Porcaro, G.; Pavone-Cossut, M.R.; Moretti, S.; Bilotta, G.; Aragona, C.; Unfer, V. Oral Treatment with EGCG, Folic Acid, Vitamin B12, and Hyaluronic Acid Improves HPV Clearance and Counteracts Its Persistence: A Clinical Study. 2025, 26, 5251. https://doi.org/10.3390/ijms26115251. 42. Weinberg M, Sar-Shalom Nahshon C, Feferkorn I, Bornstein J. Evaluation of human papilloma virus in semen as a risk factor for low sperm quality and poor in vitro fertilization outcomes: a systematic review and meta-analysis. Fertil Steril. 2020May;113(5):955-969.e4. doi: 10.1016/j.fertnstert.2020.01.010.
- [Result] Tinelli A, Gustapane S, Licchelli M, Coluccia AC, Panese G, Proietti S, Gambioli R. Treatment with Epigallocatechin Gallate, Folic Acid, Vitamin B12, and Hyaluronic Acid Decreases HPV Positivity in Women Attending Regional Screening in Puglia. Microorganisms. 2024 Sep 14;12(9):1897. doi: 10.3390/microorganisms12091897. PMID 39338571
- [Result] Aragona C, Bezerra Espinola MS, Bilotta G, Porcaro G, Calcagno M. Evaluating the Efficacy of Pervistop(R), a New Combination Based on EGCG, Folic Acid, Vitamin B12 and Hyaluronic Acid on Patients with Human Papilloma Virus (HPV) Persistent Infections and Cervical Lesions: A Pilot Study. J Clin Med. 2023 Mar 10;12(6):2171. doi: 10.3390/jcm12062171. PMID 36983172
- [Result] Ono A, Koshiyama M, Nakagawa M, Watanabe Y, Ikuta E, Seki K, Oowaki M. The Preventive Effect of Dietary Antioxidants on Cervical Cancer Development. Medicina (Kaunas). 2020 Nov 10;56(11):604. doi: 10.3390/medicina56110604. PMID 33182663
- [Result] Kwanbunjan K., Saengkar P., Cheeramakara C., Thanomsak W., Benjachai W.,Laisupasin P., Buchachart K., Songmuaeng K., Boontaveeyuwat N. Low folate status as a risk factor for cervical dysplasia in Thai women. Nutr. Res. 2005;25:641-654. doi: 10.1016/j.nutres.2005.05.004.
- [Result] Hernandez BY, McDuffie K, Wilkens LR, Kamemoto L, Goodman MT. Diet and premalignant lesions of the cervix: evidence of a protective role for folate, riboflavin, thiamin, and vitamin B12. Cancer Causes Control. 2003 Nov;14(9):859-70. doi: 10.1023/b:caco.0000003841.54413.98. PMID 14682443
- [Result] Piyathilake CJ, Henao OL, Macaluso M, Cornwell PE, Meleth S, Heimburger DC, Partridge EE. Folate is associated with the natural history of high-risk human papillomaviruses. Cancer Res. 2004 Dec 1;64(23):8788-93. doi: 10.1158/0008-5472.CAN-04-2402. PMID 15574793
- [Result] Piyathilake CJ, Macaluso M, Chambers MM, Badiga S, Siddiqui NR, Bell WC, Edberg JC, Partridge EE, Alvarez RD, Johanning GL. Folate and vitamin B12 may play a critical role in lowering the HPV 16 methylation-associated risk of developing higher grades of CIN. Cancer Prev Res (Phila). 2014 Nov;7(11):1128-37. doi: 10.1158/1940-6207.CAPR-14-0143. Epub 2014 Aug 21. PMID 25145486
- [Result] Sedjo RL, Inserra P, Abrahamsen M, Harris RB, Roe DJ, Baldwin S, Giuliano AR. Human papillomavirus persistence and nutrients involved in the methylation pathway among a cohort of young women. Cancer Epidemiol Biomarkers Prev. 2002 Apr;11(4):353-9. PMID 11927495
- [Result] Zhang D, Wen X, Wu W, Guo Y, Cui W. Elevated homocysteine level and folate deficiency associated with increased overall risk of carcinogenesis: meta-analysis of 83 case-control studies involving 35,758 individuals. PLoS One. 2015 May 18;10(5):e0123423. doi: 10.1371/journal.pone.0123423. eCollection 2015. PMID 25985325
- [Result] Ahn WS, Yoo J, Huh SW, Kim CK, Lee JM, Namkoong SE, Bae SM, Lee IP. Protective effects of green tea extracts (polyphenon E and EGCG) on human cervical lesions. Eur J Cancer Prev. 2003 Oct;12(5):383-90. doi: 10.1097/00008469-200310000-00007. PMID 14512803
- [Result] Yap JKW, Kehoe ST, Woodman CBJ, Dawson CW. The Major Constituent of Green Tea, Epigallocatechin-3-Gallate (EGCG), Inhibits the Growth of HPV18-Infected Keratinocytes by Stimulating Proteasomal Turnover of the E6 and E7 Oncoproteins. Pathogens. 2021 Apr 11;10(4):459. doi: 10.3390/pathogens10040459. PMID 33920477
- [Result] Zou C, Liu H, Feugang JM, Hao Z, Chow HH, Garcia F. Green tea compound in chemoprevention of cervical cancer. Int J Gynecol Cancer. 2010 May;20(4):617-24. doi: 10.1111/IGC.0b013e3181c7ca5c. PMID 20686382
- [Result] Chu C, Deng J, Man Y, Qu Y. Green Tea Extracts Epigallocatechin-3-gallate for Different Treatments. Biomed Res Int. 2017;2017:5615647. doi: 10.1155/2017/5615647. Epub 2017 Aug 13. PMID 28884125
- [Result] Tzellos TG, Sardeli C, Lallas A, Papazisis G, Chourdakis M, Kouvelas D. Efficacy, safety and tolerability of green tea catechins in the treatment of external anogenital warts: a systematic review and meta-analysis. J Eur Acad Dermatol Venereol. 2011 Mar;25(3):345-53. doi: 10.1111/j.1468-3083.2010.03796.x. PMID 21294779
- [Result] Tatti S, Swinehart JM, Thielert C, Tawfik H, Mescheder A, Beutner KR. Sinecatechins, a defined green tea extract, in the treatment of external anogenital warts: a randomized controlled trial. Obstet Gynecol. 2008 Jun;111(6):1371-9. doi: 10.1097/AOG.0b013e3181719b60. PMID 18515521
- [Result] Stockfleth E, Beti H, Orasan R, Grigorian F, Mescheder A, Tawfik H, Thielert C. Topical Polyphenon E in the treatment of external genital and perianal warts: a randomized controlled trial. Br J Dermatol. 2008 Jun;158(6):1329-38. doi: 10.1111/j.1365-2133.2008.08520.x. Epub 2008 Mar 20. PMID 18363746
- [Result] Gross G, Meyer KG, Pres H, Thielert C, Tawfik H, Mescheder A. A randomized, double-blind, four-arm parallel-group, placebo-controlled Phase II/III study to investigate the clinical efficacy of two galenic formulations of Polyphenon E in the treatment of external genital warts. J Eur Acad Dermatol Venereol. 2007 Nov;21(10):1404-12. doi: 10.1111/j.1468-3083.2007.02441.x. PMID 17958849
- [Result] Fiorillo L, Cervino G, Surace G, De Stefano R, Laino L, D'Amico C, Fiorillo MT, Meto A, Herford AS, Arzukanyan AV, Spagnuolo G, Cicciu M. Human Papilloma Virus: Current Knowledge and Focus on Oral Health. Biomed Res Int. 2021 Feb 1;2021:6631757. doi: 10.1155/2021/6631757. eCollection 2021. PMID 33623784
- [Result] Pal A, Kundu R. Human Papillomavirus E6 and E7: The Cervical Cancer Hallmarks and Targets for Therapy. Front Microbiol. 2020 Jan 21;10:3116. doi: 10.3389/fmicb.2019.03116. eCollection 2019. PMID 32038557
- [Result] Kato Y, Shigehara K, Nakagawa T, Nakata H, Iijima M, Nakashima K, Kawaguchi S, Izumi K, Kadono Y, Mizokami A. Human papillomavirus detected in sperm of Japanese infertile males affects reproductive parameters. Int J Infect Dis. 2021 Nov;112:294-299. doi: 10.1016/j.ijid.2021.09.029. Epub 2021 Sep 20. PMID 34547493
- [Result] Schillaci R, Capra G, Bellavia C, Ruvolo G, Scazzone C, Venezia R, Perino A. Detection of oncogenic human papillomavirus genotypes on spermatozoa from male partners of infertile couples. Fertil Steril. 2013 Nov;100(5):1236-40. doi: 10.1016/j.fertnstert.2013.06.042. Epub 2013 Jul 24. PMID 23891022
- [Result] De Toni L, Muscianisi F, Corsini C, Ghezzi M, Di Nisio A, Foresta C, Garolla A. Serum Anti-HPV Antibody Titer as a Marker of Vaccine Effectiveness in Males with Genital Infection. Vaccines (Basel). 2020 Dec 7;8(4):743. doi: 10.3390/vaccines8040743. PMID 33297367
- [Result] Foresta C, Noventa M, De Toni L, Gizzo S, Garolla A. HPV-DNA sperm infection and infertility: from a systematic literature review to a possible clinical management proposal. Andrology. 2015 Mar;3(2):163-73. doi: 10.1111/andr.284. Epub 2014 Oct 1. PMID 25270519
- [Result] Foresta C, Garolla A, Zuccarello D, Pizzol D, Moretti A, Barzon L, Palu G. Human papillomavirus found in sperm head of young adult males affects the progressive motility. Fertil Steril. 2010 Feb;93(3):802-6. doi: 10.1016/j.fertnstert.2008.10.050. Epub 2008 Dec 18. PMID 19100537
- [Result] Lenzi A, Mirone V, Gentile V, Bartoletti R, Ficarra V, Foresta C, Mariani L, Mazzoli S, Parisi SG, Perino A, Picardo M, Zotti CM. Rome Consensus Conference - statement; human papilloma virus diseases in males. BMC Public Health. 2013 Feb 7;13:117. doi: 10.1186/1471-2458-13-117. PMID 23391351
- [Result] Laprise C, Trottier H, Monnier P, Coutlee F, Mayrand MH. Prevalence of human papillomaviruses in semen: a systematic review and meta-analysis. Hum Reprod. 2014 Apr;29(4):640-51. doi: 10.1093/humrep/det453. Epub 2013 Dec 22. PMID 24365799
- [Result] Perez-Andino J, Buck CB, Ribbeck K. Adsorption of human papillomavirus 16 to live human sperm. PLoS One. 2009 Jun 9;4(6):e5847. doi: 10.1371/journal.pone.0005847. PMID 19513123
- [Result] Zacharis K, Messini CI, Anifandis G, Koukoulis G, Satra M, Daponte A. Human Papilloma Virus (HPV) and Fertilization: A Mini Review. Medicina (Kaunas). 2018 Jul 27;54(4):50. doi: 10.3390/medicina54040050. PMID 30344281
- [Result] Garolla A, Engl B, Pizzol D, Ghezzi M, Bertoldo A, Bottacin A, Noventa M, Foresta C. Spontaneous fertility and in vitro fertilization outcome: new evidence of human papillomavirus sperm infection. Fertil Steril. 2016 Jan;105(1):65-72.e1. doi: 10.1016/j.fertnstert.2015.09.018. Epub 2015 Oct 9. PMID 26453270
- [Result] Lorenzon L, Terrenato I, Dona MG, Ronchetti L, Rollo F, Marandino F, Carosi M, Diodoro MG, Sentinelli S, Visca P, Vocaturo G, Bellardini P, Vocaturo A, Benevolo M. Prevalence of HPV infection among clinically healthy Italian males and genotype concordance between stable sexual partners. J Clin Virol. 2014 Jul;60(3):264-9. doi: 10.1016/j.jcv.2014.04.003. Epub 2014 Apr 15. PMID 24794396
- [Result] Kero K, Rautava J. HPV Infections in Heterosexual Couples: Mechanisms and Covariates of Virus Transmission. Acta Cytol. 2019;63(2):143-147. doi: 10.1159/000494710. Epub 2019 Feb 22. PMID 30799413
- [Result] Widdice L, Ma Y, Jonte J, Farhat S, Breland D, Shiboski S, Moscicki AB. Concordance and transmission of human papillomavirus within heterosexual couples observed over short intervals. J Infect Dis. 2013 Apr 15;207(8):1286-94. doi: 10.1093/infdis/jit018. Epub 2013 Jan 14. PMID 23319742
- [Result] Giuliano AR, Nyitray AG, Kreimer AR, Pierce Campbell CM, Goodman MT, Sudenga SL, Monsonego J, Franceschi S. EUROGIN 2014 roadmap: differences in human papillomavirus infection natural history, transmission and human papillomavirus-related cancer incidence by gender and anatomic site of infection. Int J Cancer. 2015 Jun 15;136(12):2752-60. doi: 10.1002/ijc.29082. Epub 2014 Jul 26. PMID 25043222
- [Result] de Sanjose S, Serrano B, Castellsague X, Brotons M, Munoz J, Bruni L, Bosch FX. Human papillomavirus (HPV) and related cancers in the Global Alliance for Vaccines and Immunization (GAVI) countries. A WHO/ICO HPV Information Centre Report. Vaccine. 2012 Nov 20;30 Suppl 4:D1-83, vi. doi: 10.1016/S0264-410X(12)01435-1. No abstract available. PMID 23510764
- [Result] Doorbar J, Quint W, Banks L, Bravo IG, Stoler M, Broker TR, Stanley MA. The biology and life-cycle of human papillomaviruses. Vaccine. 2012 Nov 20;30 Suppl 5:F55-70. doi: 10.1016/j.vaccine.2012.06.083. PMID 23199966
- [Result] Cid Arregui A, Gariglio P, Kanda T, Doorbar J. ONCOGENIC HUMAN PAPILLOMAVIRUSES: High-Risk Human Papillomaviruses: Towards a Better Understanding of the Mechanisms of Viral Transformation, Latency and Immune-Escape. Open Virol J. 2012;6:160-2. doi: 10.2174/1874357901206010160. Epub 2012 Dec 28. No abstract available. PMID 23346264
- [Result] McLaughlin-Drubin ME, Munger K. Oncogenic activities of human papillomaviruses. Virus Res. 2009 Aug;143(2):195-208. doi: 10.1016/j.virusres.2009.06.008. Epub 2009 Jun 18. PMID 19540281
- [Result] Bosch FX, Broker TR, Forman D, Moscicki AB, Gillison ML, Doorbar J, Stern PL, Stanley M, Arbyn M, Poljak M, Cuzick J, Castle PE, Schiller JT, Markowitz LE, Fisher WA, Canfell K, Denny LA, Franco EL, Steben M, Kane MA, Schiffman M, Meijer CJ, Sankaranarayanan R, Castellsague X, Kim JJ, Brotons M, Alemany L, Albero G, Diaz M, de Sanjose S; ICO Monograph 'Comprehensive Control of HPV Infections and Related Diseases' Vaccine Volume 30, Supplement 5, 2012. Comprehensive control of human papillomavirus infections and related diseases. Vaccine. 2013 Dec 30;31 Suppl 6:G1-31. doi: 10.1016/j.vaccine.2013.10.002. PMID 24331817
- [Result] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338